CLINICAL TRIAL: NCT06148857
Title: Prevalence Data for Total Corneal Astigmatism in Cataract Surgery Candidates
Brief Title: Total Corneal Astigmatism Prevalence in Cataract Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BLB2
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cataract
Keywords: cataract; astigmatism; prevalence
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IOLMaster 700 — The IOLMaster 700, one of the most commonly used optical biometers for IOL power calculation, measures the anterior corneal surface radius using a telecentric keratometry. Additionally, it employs swept-source optical coherence tomography (SS-OCT) technology to simultaneously measures the posterior cornea surface radius and central corneal thickness (CCT).
  The AK formula, described by Abulafia et al., is a regression formula that calculates an estimated TCA using K astigmatism.
  The Barrett toric calculator uses an unpublished mathematical prediction method of TCA based on anterior corneal measurements.
  Other Names: the Abulafia-Koch formula; the Barrett toric calculator

SUMMARY:
The purpose of this study is to report the prevalence data for total corneal astigmatism (TCA) in cataract surgery candidates.

DETAILED DESCRIPTION:
The purpose of this retrospective study is to report the prevalence data for total corneal astigmatism (TCA) in cataract surgery candidates. Preoperative biometric data of all the patients who underwent cataract surgery in the Department of Ophthalmology, Peking University Third Hospital, from January 2019 to May 2023, were collected and analyzed. Data sets with incomplete biometric data were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cataract surgery in the Department of Ophthalmology, Peking University Third Hospital from January 2019 to May 2023.

Exclusion Criteria:

* Incomplete biometric data .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who underwent cataract surgery in the Department of Ophthalmology, Peking University Third Hospital from January 2019 to May 2023.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
total keratometric astigmatism | At Enrollment
  Total keratometry is calculated based on the anterior and posterior corneal surface radius and CCT using the thick lens formula with the actual indices of refractions for air (1.000), cornea (1.376), and aqueous (1.336) by IOLMaster 700. Total keratometric astigmatism is taken as the TCA measured by IOLMaster 700.
Abulafia-Koch formula total corneal astigmatism | At Enrollment
  The AK formula, described by Abulafia et al, is a regression formula that calculates an estimated TCA using K astigmatism.
Barrett toric calculator total corneal astigmatism | At Enrollment
  The Barrett toric calculator uses an unpublished mathematical prediction method of TCA based on anterior corneal measurements. AL, ACD, LT, WTW, and K data by IOLMaster 700 were input into the Barrett toric calculator. The target refraction, incision surgically induced astigmatism (SIA), and incision location were all set as 0. The output net astigmatism was recorded as TCA predicted by the Barrett toric calculator.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No